CLINICAL TRIAL: NCT03131843
Title: A Pilot Randomized Controlled Trial Assessing the Effectiveness of Alcohol Swabs in Preventing Infections in Pediatric Patients Receiving Vaccinations
Brief Title: Effectiveness of Alcohol Swabs for Preventing Infections During Vaccination
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Anna Taddio, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 33391
Record Dates: First submitted 2017-04-17; First posted 2017-04-27 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Skin Infection
Keywords: skin infection; vaccination; children; alcohol swab; skin preparation
MeSH Terms: conditions — Cellulitis | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, parents, care providers and outcomes assessors will not be aware of whether the participant was swabbed in the location of the vaccine injection. Only the investigator will know where alcohol was applied on the skin relative to the vaccine injection site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol (Experimental): Alcohol will be wiped on the vaccine injection site immediately before vaccine injection.
  Interventions: Drug: Alcohol
- No alcohol (Placebo Comparator): Alcohol will be wiped adjacent to the vaccine injection site immediately before vaccine injection.
  Interventions: Drug: No alcohol

INTERVENTIONS:
Drug: Alcohol — Alcohol cleansing swab/wipe
  Arms: Alcohol
Drug: No alcohol — No alcohol will be used; alcohol cleansing swab/wipe will be used at a different injection site
  Arms: No alcohol

SUMMARY:
Alcohol is used to disinfect the skin prior to injections in order to prevent infections caused by bacteria on the skin being injected within tissue. At present, however, clinical trials do not demonstrate a clinical impact of using or not using alcohol swabs on infections and infection symptoms calling into question the practice of using it prior to all injections. These studies are methodologically flawed, and do not specifically examine vaccine injections. The present study is being undertaken to provide some preliminary data for the risk of infection and infection symptoms when alcohol swabs are not used to perform vaccine injections.

DETAILED DESCRIPTION:
Alcohol is used to disinfect the skin prior to injections in order to prevent infections caused by bacteria on the skin being injected within tissue. Alcohol has been shown to be a good disinfectant, reducing the number of bacteria on skin by 47-91%. However, in previous clinical trials, there has been no clinical impact of using or not using alcohol swabs on infections and infection symptoms calling into question the practice of using it prior to all injections. These studies, however, are generally of low scientific rigor (e.g., not randomized, not blinded, did not use standard case definitions of the adverse reactions being measured). Moreover, it is important to note that none of them specifically evaluated vaccine injections, the most common type of injection worldwide.

At present, based on the available evidence base, the World Health Organization (WHO) and the Centre for Disease Control (CDC) do not recommend the use of alcohol swabs before vaccine injections. As a result, immunizers in many countries around the world currently do not cleanse the skin with alcohol prior to vaccination. Despite these recommendations, clinicians in our community and across Canada commonly use alcohol swabs prior to all vaccine injections. In this application, investigators will undertake a pilot randomized study to evaluate the incidence of infection symptoms and infections in children undergoing vaccination with and without skin cleansing with alcohol swabs.

ELIGIBILITY:
Inclusion Criteria:

* healthy pediatric patients undergoing routine vaccinations

Exclusion Criteria:

* no contra-indications to vaccination or alcohol swab,
* ability to understand English and consent to the study

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 170 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Skin infection | within 14 days of injection
  skin infection (cellulitis, abscess), defined as per Brighton Collaboration definition (2007)

SECONDARY OUTCOMES:
Skin infection symptoms | within 14 days of injection
  skin infection symptoms (redness, swelling, pain, warmth, discharge), defined as per Brighton Collaboration definition (2007)
Feasibility of recruitment | from date of first enrollment until the date of final enrollment, up to 1 year
  recruitment rate for study
Compliance with protocol | within 30 days of injection
  rate of parent compliance with study procedures
Feasibility of protocol | from the date of first enrollment until the date of the last follow-up, or study completion, up to 1 year
  descriptives of adverse events relative to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — University of Toronto
Locations (1):
- Pediatrician Clinic, North York, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.